CLINICAL TRIAL: NCT00541957
Title: Randomized Trial of Psychotherapy for Persistently Depressed Primary Care Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Memorial Hospital of Rhode Island (Other)
Responsible Party: Lisa Uebelacker, Ph.D., PI, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH067779 (NIH)
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Major Depression
Keywords: Major depression; Primary care
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Other): Medication prescribed by PCP
  Interventions: Drug: Medication prescribed by PCP
- 1 (Experimental): Medication prescribed by PCP + behavior therapy
  Interventions: Behavioral: behavior therapy; Drug: Medication prescribed by PCP

INTERVENTIONS:
Behavioral: behavior therapy — 10 sessions over 4 months
  Arms: 1
Drug: Medication prescribed by PCP — Can include any antidepressant medication

SUMMARY:
This is a pilot study. The purpose of this study is to determine whether adding 4 months of behavioral therapy to primary care physician medication treatment(relative to medication treatment alone) improves outcomes for persistently depressed primary care patients.

ELIGIBILITY:
Inclusion Criteria:

* Current MDD or MDD within the past year or current dysthymia
* PHQ-9 > 10
* have been prescribed an antidepressant medication (by their PCP) at least 8 weeks before pre-treatment timepoint
* are able to speak, read, and understand English sufficiently well to complete study procedures
* are between the ages of 18 and 70

Exclusion Criteria:

* presence of significant suicidal ideation or risk
* history of bipolar disorder, schizophrenia, psychotic symptoms, or severe alcohol or drug problems within the past year;
* history of antisocial personality disorder or borderline personality disorder;
* currently in psychotherapy or have received counseling more frequently than once per month in the past year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Depression symptoms | 4 months

SECONDARY OUTCOMES:
Psychosocial functioning | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital
Locations (2):
- United States (2):
  - Memorial Hospital of RI, Pawtucket, Rhode Island
  - Butler Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Uebelacker LA, German NM, Gaudiano BA, Miller IW. Patient health questionnaire depression scale as a suicide screening instrument in depressed primary care patients: a cross-sectional study. Prim Care Companion CNS Disord. 2011;13(1):PCC.10m01027. doi: 10.4088/PCC.10m01027. PMID 21731830